CLINICAL TRIAL: NCT04816591
Title: Middle Meningeal Artery Embolization for the Treatment of Subdural Hematomas With TRUFILL® n-BCA
Acronym: MEMBRANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNV_2020_01
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma, MMA Embolization
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Experimental: Interventional Cohort: Treatment Arm (Experimental): Standard of Care Surgery + Embolization
  Interventions: Device: Experimental: Interventional Cohort: TRUFILL n-Butyl Cyanoacrylate (n-BCA) Liquid Embolic System
- Standard of Care Surgery Only (Active Comparator): Standard of Care Surgery Only
  Interventions: Other: Standard of Care Surgery
- Interventional Cohort: Treatment Arm (Experimental): Standard of Care Medical Management + Embolization
  Interventions: Device: Experimental: Interventional Cohort: TRUFILL n-BCA Liquid Embolic System
- Standard of Care Medical Management Only (Active Comparator): Standard of Care medical management only.
  Interventions: Other: Standard of Care Medical Management

INTERVENTIONS:
Device: Experimental: Interventional Cohort: TRUFILL n-Butyl Cyanoacrylate (n-BCA) Liquid Embolic System — Standard of Care Surgery + Embolization
  Arms: Experimental: Interventional Cohort: Treatment Arm
Other: Standard of Care Surgery — Standard of Care Surgery Only
  Arms: Standard of Care Surgery Only
Device: Experimental: Interventional Cohort: TRUFILL n-BCA Liquid Embolic System — Standard of Care Medical Management + Embolization
  Arms: Interventional Cohort: Treatment Arm
Other: Standard of Care Medical Management — Standard of Care Medical Management Only
  Arms: Standard of Care Medical Management Only

SUMMARY:
This is a prospective, multi-center, open-label, randomized controlled study in which subjects can receive standard of care (SOC) alone or SOC and TRUFILL n-BCA MMA embolization for the treatment of chronic subdural hematomas (cSDH).

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, randomized controlled study in which up to 376 subjects will be randomized to receive standard of care (SOC) alone or SOC and TRUFILL n-BCA MMA embolization for the treatment of cSDH.

ELIGIBILITY:
Inclusion Criteria:

* Pre-randomization mRS </= 3
* Confirmed diagnosis of chronic subdural hematoma
* Completed informed consent

Exclusion Criteria:

* Acute subdural hematoma
* Prior treatment of target subdural hematoma
* Markwalder assessment >/= 3
* Glasgow Coma Scale < 9
* Presumed microbial superinfection
* CT or MRI evidence of intracranial tumor or mass lesion
* Life expectancy < 1 year
* Women who are pregnant, lactating, or who are of childbearing age and plan on becoming pregnant during the study
* Current involvement in another clinical trial that may confound study endpoints

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Effectiveness | 180 days post procedure
  Hematoma recurrence/progression or requiring re-intervention
Occurrence of All Adverse Events (AEs) up to 6 Months | Up to 6 months
  AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated.

SECONDARY OUTCOMES:
Effectiveness | 180 days post procedure
  Reduction of hematoma volume
Safety: Change in mRS | 180 days post procedure
  Change in mRS

OTHER OUTCOMES:
Health Economics | 365 days post procedure
  Hospital days

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kellner, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Ansaar Rai, MD, Principal Investigator — West Virginia University
Locations (33):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Carondelet St Joseph's Hospital, Tucson, Arizona
  - John Muir Physician Network Clinical Research Center, Walnut Creek, California
  - Swedish Medical Center, Englewood, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - Baptist Medical Center, Jacksonville, Florida
  - University of Miami - Jackson Memorial Hospital, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Wellstar Health System, Marietta, Georgia
  - Memorial Health University Health Center, Savannah, Georgia
  - University of Maryland, Baltimore, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio Health, Columbus, Ohio
  - Mercy Health St Vincent Medical Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital of Research, Pittsburgh, Pennsylvania
  - Semmes Murphey Foundation, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Stroke Institute, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - West Virginia Hospital, Morgantown, West Virginia
- China (2):
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu.

REFERENCES:
- [Derived] Kellner CP, Al-Mufti F, Gupta R, Jankowitz BT, Starke RM, Rai AT. Middle Meningeal Artery Embolization with n-Butyl Cyanoacrylate for the Treatment of Subdural Hematomas: The MEMBRANE Study Design. Stroke Vasc Interv Neurol. 2025 Sep 17;5(6):e001828. doi: 10.1161/SVIN.125.001828. eCollection 2025 Nov. PMID 41608724